CLINICAL TRIAL: NCT02506088
Title: Preventing Sexual Aggression Among High School Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Lindsay Orchowski Ph.D., Staff Psychologist, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1U01CE002531 (NIH)
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Your Voice Your View (Experimental): Participants in schools assigned to the treatment group will engage in a four session intervention aimed at prevention of sexual violence. Your Voice Your View is grounded in social norms theory and bystander intervention training. The intervention also includes a social norms marketing campaign.
  Interventions: Behavioral: Your Voice Your View
- Wait List Control Group (No Intervention): Participants in schools assigned to the wait list control group will complete survey assessments at the same schedule as schools assigned to the treatment group. Schools will have the option to implement Your Voice Your View following completion of the 6-month survey.

INTERVENTIONS:
Behavioral: Your Voice Your View — Session 1 of the intervention involves background information, an introduction to social norms, and bystander intervention skills training. Session 2 of the intervention establishes conditions for consent, types of abusive behavior and identifying abuse. Session 3 of the intervention addresses risk reduction strategies for girls. Session 3 of the intervention addresses false accusations, masculinity, and additional practice on identifying conditions for consent for boys. Session 4 of the intervention includes active practice of bystander intervention skills.
  Arms: Your Voice Your View

SUMMARY:
The present research creates a partnership between researchers and a community agency to evaluate whether a sexual assault prevention program for high school students reduces perpetration of sexual violence among high school boys.

DETAILED DESCRIPTION:
The present research advances the science of sexual assault prevention by creating a mutually beneficial partnership between well-established sexual assault prevention researchers and a CDC Rape Prevention and Education Program (RPE)-funded community agency to conduct a rigorous experimental evaluation of universal primary prevention programming designed to reduce sexual aggression among high school boys. The present research tests multi-session prevention programming that targets change at multiple levels of the social ecology (i.e., individual-, peer- and community-level) through social norms theory and bystander education. Specifically, the present research evaluates Your Voice Your View. Your Voice Your View was developed and is currently administered in Rhode Island High Schools by the CDC RPE-funded agency Day One of Rhode Island. The program will be tested in a group randomized cluster trial among 10th graders at 30 high schools, with the aim of reducing perpetration of sexual aggression among high school boys.

Specifically, this research will conduct a randomized controlled trial with a sample of 10th grade students to demonstrate efficacy of the intervention in reducing rates of sexual aggression among high school boys, rates of dating violence involvement, and related risk and protective factors over a 2- and 6-month follow-up in comparison to a wait-list control group. Thirty schools will be matched on demographic characteristics (i.e., % receiving subsidized lunch, racial/ethnic minority enrollment) and randomized to receive Your Voice Your View or to the wait-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents at Rhode Island high schools will be eligible for enrollment according to the following criteria: 1) adolescent assent given; 3) passive consent of a parent/legal guardian is given. Teachers will be eligible to participate in educator assessments if consent is given.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7910 (Actual)
Dates: Start 2015-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Perpetration of Sexual Violence Survey | up to 6-months

SECONDARY OUTCOMES:
Rate of Dating Violence Perpetration | up to 6 months
Rape Myth Acceptance Survey | up to 6 months
Bystander Intervention Skills Survey | up to 6 months
  Composite measure: Increase Positive Bystander Behavior, Decrease Barriers to Intervening, Increase Likelihood of Intervening

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay M. Orchowski, Ph.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States